CLINICAL TRIAL: NCT06320028
Title: Altering Default Mode Network Activity to Reduce Depressive Symptoms
Brief Title: Altering Default Mode Network Activity With Transcranial Focused Ultrasound to Reduce Depressive Symptoms
Acronym: DMNtFUS
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Openwater (Unknown)
Responsible Party: Principal Investigator, John Allen, Distinguished Professor of Psychology, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 019782-00001
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Depressive Disorder, Major; Depression
Keywords: Non-invasive Transcranial Focused Ultrasound Stimulation; Depression; Mood disorders
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Mood Disorders

STUDY DESIGN:
Intervention Model Description: All participants will receive the same treatment protocol.
Masking Description: There is no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-invasive Transcranial Focused Ultrasound (Experimental): Device: Transcranial Ultrasound Power
  The ultrasound will be delivered using a custom Neuromodulation device consisting of 128 element ultrasound array (Openwater) with the ultrasound beam having the following parameters: acoustic frequency = 400 kHz, pulse duration = 5 ms, pulse repetition rate (PRR) = 10 Hz, spatial peak/temporal average acoustic intensity = 435 mW /cm2, peak negative pressure 650 kPa. The ultrasound probe will be secured by a custom-designed headset created by Openwater. The Localite Neuronavigation Software (TMS Navigator 3.3 adapted for ultrasound device), including a 3D camera, fiducial markers on the headset and pointer, and software will register the position of the probe with respect to the patient's structural MRI.
  Interventions: Device: Non-Invasive Transcranial Focused Ultrasound

INTERVENTIONS:
Device: Non-Invasive Transcranial Focused Ultrasound — The ultrasound will be delivered for 10 minutes per treatment session targeting to the participant's amPFC.

SUMMARY:
Depression is a leading cause of disability worldwide, affecting roughly 21 million adults. Repetitive Negative Thought (RNT) has been identified as a potential maintaining factor in depression, such that those who exhibit higher degrees of RNT endorse greater symptoms. Research also suggests that the Default Mode Network (DMN), responsible for self-referential processing, plays an important role in depression wherein it has been linked to RNT. In depressed individuals, this network appears to be hyper-connected, or "too connected", within itself which, in turn, is thought to promote RNT.

Half of depressed individuals are treatment-resistant, creating a critical need to identify more effective interventions derived from a better mechanistic understanding of the development and maintenance of depression. Non-invasive Transcranial-Focused Ultrasound Stimulation (tFUS) is promising for the treatment of depression. tFUS directs a low-intensity (nonthermal) focused ultrasound beam that passes safely through the skull. Compared to other noninvasive neuromodulation approaches, tFUS can target deeper brain regions with high spatial precision.

The present study is an exploratory non-blinded single treatment study to investigate whether tFUS targeting a major hub of the DMN, the anterior-medial prefrontal cortex, can improve depression symptoms and reduce RNT. Twenty depressed individuals with high RNT (75th percentile) will complete up to eleven ultrasound sessions targeting the anterior medial prefrontal cortex, a hub of the brain's default mode network that has been found to be hyper-connected in depression. MRI scans will be obtained before the first and after the last ultrasound sessions. Based on previous literature, it is predicted that depression interview ratings and self-report symptoms will decrease after the intervention, and also that DMN connectivity will decrease following intervention.

DETAILED DESCRIPTION:
Participants will first complete the online screening to identify those who may meet criteria of major depressive disorder and have high RNT. Those meeting these criteria will be contacted for a formal diagnostic interview, consisting of the consent process and a structured clinical interview using the DSM-5. Once deemed eligible, participants will complete baseline interviews, self-report surveys, and an MRI session. Then, they will complete up to three weeks of ultrasound treatment, wherein the first week consists of five ultrasound sessions. Upon completion of week one, participants will complete the same interview, self-report surveys, and MRI session. Participants' symptom improvement will be determined by whether they meet remission criteria, defined as a Beck Depression Inventory Score - II (BDI-II) of <13 and a Hamilton Depression Rating Scale (HDRS) score of <8. If remission criteria are not met, participants will continue ultrasound sessions for two more weeks, three sessions per week. Following completion, participants will complete a final interview, self-report surveys, and MRI session. In each treatment session, the ultrasound device will be placed on the participants' forehead with the aid of the customized headset co-localized to the participant's structural MR image. Each ultrasound treatment lasts ten minutes.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 18-50
* Participants must have normal or corrected vision (glasses, contacts, etc)
* Must be proficient in English in order to read the consent form (Spanish speakers are included, as long as they are also proficient in English)
* Must be right-handed
* Upper 25% of distribution on perseverative thinking scores based on local norms (score ≥ 37)
* Participants meeting DSM-5 criteria for current major depressive episode

Participants may be excluded from the MRI portion of the experiment if they are pregnant or are unsure if they may be pregnant or have any contraindications for MRI, including severe claustrophobia, non-MRI compatible cardiac pacemakers; implantable defibrillators; aneurysm clips; neural stimulators; artificial heart valves; ear implants; insulin pumps; drug infusion devices; IUDs; magnetic dental appliances; metal fragments or foreign objects in the eyes, skin or body; metal plates, screws, and prosthetics; non-removable metal piercings; tattoos on the head and neck, other certain older tattoos or permanent makeup (eyeliner) using metal-containing inks, some medicated patches, or any other condition, metal implant or other injury or device that is contraindicated for MRI. If a subject has any of these, the experimenter will evaluate whether it is safe for them to participate in the MRI portion of the experiment.

Exclusion Criteria:

* History of head injury with loss of consciousness for more than 5 min
* Uncorrected hearing or vision impairment severe enough to interfere with participation.
* Currently have or history of brain or mental illness judged likely to interfere with testing, including drug and/or alcohol dependence
* Sleep disorder (e.g., insomnia)
* Current drug, alcohol, or prescription drug intoxication
* History of epilepsy
* History of diagnosed migraines
* Metal implants in their head or face, including dental retainers that cannot be removed
* History of cardiac problems that could impact brain function (e.g., atrial fibrillation)
* Current active suicidal potential necessitating immediate treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-06-03 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory - II (BDI-II) | Before ultrasound treatment, daily after each ultrasound session, after completion of week 1 of treatment, after completion of week 3 of treatment (if applicable)
  The BDI-II is one of the most widely used self-report measures for assessing depression. It includes 21 self-report items. Scores range from 0 to 63, and higher scores indicate higher levels of depressive symptoms. In this study, the BDI-II was used to monitor depressive symptoms over the course of treatment. In our research, we will employ the BDI-II to track changes in self-reported depressive symptoms throughout the intervention, comparing the total BDI-II scores at different assessment points to analyze the efficacy of the treatment.
Perseverative Thinking Questionnaire (PTQ) | Before ultrasound treatment, daily after each ultrasound session, after completion of week 1 of treatment, after completion of week 3 of treatment (if applicable)
  The PTQ is a commonly used self-report measure for assessing a characteristic of depression, repetitive negative thought (RNT). It includes 15 self-report items. Scores range from 0 to 60, and higher scores indicate higher levels of RNT. In this study, the PTQ was used to monitor RNT over the course of treatment. In our research, we will employ the PTQ to track changes in RNT throughout the intervention, comparing the total PTQ scores at different assessment points to analyze the efficacy of the treatment.
Hamilton Depression Rating Scale (HDRS) | Before ultrasound treatment, after completion of week 1 of treatment, after completion of week 3 of treatment (if applicable)
  The Hamilton Depression Rating Scale (HDRS) is a widely utilized clinician-administered assessment tool designed to measure the severity of depressive symptoms in individuals. Comprising 17 items, the HDRS evaluates various aspects of depression. Scores range from 0 to 52, and higher total scores indicate greater depressive symptoms. In our research, we will employ the HDRS to track changes in depressive symptoms throughout the intervention, comparing the total HDRS scores at each main time point to analyze the efficacy of the treatment.
Default Mode Network (DMN) Connectivity | Before ultrasound treatment, after completion of week 1 of treatment, after completion of week 3 of treatment (if applicable)
  The DMN is a set of brain regions known to be "hyperconnected" in depressed individuals and may be a potential biomarker for this costly disorder. In our research, we will compare DMN connectivity at each major time point to observe whether there is a decrease in DMN connectivity to assess the efficacy of treatment.

SECONDARY OUTCOMES:
The Montgomery-Åsberg Depression Rating Scale (MADRS) | Before ultrasound treatment, after completion of week 1 of treatment, after completion of week 3 of treatment (if applicable)
  The MADRS is a clinician-administered assessment tool commonly used to evaluate the severity of depressive symptoms in individuals. It consists of 10 items that assess various aspects of depression. Scores range from 0 to 60, with higher scores indicating more severe depressive symptoms. In our research, we will employ the MADRS to track changes in depressive symptoms throughout the intervention, comparing the total MADRS scores at each main time point to analyze the efficacy of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John JB Allen, PhD, Principal Investigator — University of Arizona Psychology Department; Jessica N Schachtner, BA, Principal Investigator — University of Arizona Psychology Department
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fini M, Tyler WJ. Transcranial focused ultrasound: a new tool for non-invasive neuromodulation. Int Rev Psychiatry. 2017 Apr;29(2):168-177. doi: 10.1080/09540261.2017.1302924. Epub 2017 Apr 21. PMID 28430535
- [Background] Kubanek J. Neuromodulation with transcranial focused ultrasound. Neurosurg Focus. 2018 Feb;44(2):E14. doi: 10.3171/2017.11.FOCUS17621. PMID 29385924
- [Background] Samantha J. Reznik, Joseph L. Sanguinetti, William J. Tyler, Chris Daft, John J.B. Allen. (2020) A double-blind pilot study of transcranial ultrasound (TUS) as a five-day intervention: TUS mitigates worry among depressed participants, Neurology, Psychiatry and Brain Research, 37(60-66), ISSN 0941-9500, https://doi.org/10.1016/j.npbr.2020.06.004.
- [Background] Sanguinetti JL, Hameroff S, Smith EE, Sato T, Daft CMW, Tyler WJ, Allen JJB. Transcranial Focused Ultrasound to the Right Prefrontal Cortex Improves Mood and Alters Functional Connectivity in Humans. Front Hum Neurosci. 2020 Feb 28;14:52. doi: 10.3389/fnhum.2020.00052. eCollection 2020. PMID 32184714
- [Background] Sanguinetti, J. L., Smith, E., Allen, J. J. B., Hameroff, S. (2014). Human brain stimulation with transcranial ultrasound (TUS); Potential applications for mental health. In Bioelectromagnetic Medicine. New York, NY: Taylor & Francis.
- [Background] Sheline YI, Barch DM, Price JL, Rundle MM, Vaishnavi SN, Snyder AZ, Mintun MA, Wang S, Coalson RS, Raichle ME. The default mode network and self-referential processes in depression. Proc Natl Acad Sci U S A. 2009 Feb 10;106(6):1942-7. doi: 10.1073/pnas.0812686106. Epub 2009 Jan 26. PMID 19171889
- [Derived] Schachtner JN, Dahill-Fuchel JF, Zhang D, Allen KE, Bawiec CR, Hollender PJ, Ornellas SB, Konecky SD, Achrol AS, Allen JJB. The effect of non-invasive transcranial focused ultrasound for depression on the default mode network: an open-label pilot trial. Front Psychiatry. 2026 Jan 20;16:1722575. doi: 10.3389/fpsyt.2025.1722575. eCollection 2025. PMID 41641082
- [Derived] Schachtner JN, Dahill-Fuchel JF, Allen KE, Bawiec CR, Hollender PJ, Ornellas SB, Konecky SD, Achrol AS, Allen JJB. Transcranial focused ultrasound targeting the default mode network for the treatment of depression. Front Psychiatry. 2025 Apr 4;16:1451828. doi: 10.3389/fpsyt.2025.1451828. eCollection 2025. PMID 40256163

DOCUMENTS (2):
  • Statistical Analysis Plan (2024-01-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT06320028/SAP_000.pdf
  • Informed Consent Form (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT06320028/ICF_001.pdf